CLINICAL TRIAL: NCT03834051
Title: Prospective, Open-label Trial to Evaluate Efficacy of Fecal Microbiota Transplantation for Treatment of Chronic Gastrointestinal Dysbiosis or Clearance of Antimicrobial Resistant Organism.
Brief Title: Fecal Microbiota Transplantation for Treatment of Gastrointestinal Dysbiosis or Clearance of ARO
Acronym: FMTGID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vancouver Island Health Authority (Other)
Responsible Party: Principal Investigator, Christine Lee, MD, Vancouver Island Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GID.FMT
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2023-08

CONDITIONS: Dysbiosis; Antimicrobial Resistant Organism
MeSH Terms: conditions — Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Fecal Microbiota Transplantation
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation Rectal Administration Open Label

SUMMARY:
The objective of this study is to assess the efficacy of FMTs via rectal administration for 1) symptom improvement in individuals with a formal diagnosis of dysbiosis due to active inflammatory bowel disease or irritable bowel syndrome; 2) clearance of antimicrobial resistant organism from the gastrointestinal tract.

DETAILED DESCRIPTION:
Fecal Microbiota Transplantation (FMT), which had been predominantly utilized by the veterinarians until late 1990's has generated a significant interest for its potential use in various gastrointestinal, psychiatric, neurologic and metabolic disorders within the past few years. Since 2010, there has been an explosion of research, publications and media coverage related to the high efficacy range, 80 - 90% for treatment of recurrent Clostridioides (Clostridium) difficile infection (rCDI). The exact mechanisms of its success in curing CDI are yet to be discovered. Metagenomic studies have shown that patients with rCDI lack protective and diverse colonic microbiome and remain in a state of chronic dysbiosis. Following a successful FMT, the microbiome of a patient with rCDI resembles that of the donor's and remains as such overtime. There is no precise and agreed definition of dysbiosis. For the purpose of this study, dysbiosis is defined as perturbation of host-microbial interactions which results in compositional changes in the fecal microbiota as determined by clinical criteria of constellation of symptoms, including change in the bowel function (diarrhea, constipation or bloating) in which an alteration of the microbiota is either known based on molecular or culture-based profiling or suspected according to the history, which includes but is not limited to repeated or prolonged use of antibiotics or gastrointestinal infection.

The cause of inflammatory bowel dieseases (IBD) is unknown but studies have shown that IBD is a chronic inflammatory disease with altered and decreased microbiota diversity of the gastrointestinal tract when compared to the healthy individuals. Canada has the highest incidence of IBD in the world. The annual total (direct and indirect) health costs is estimated to $2.8 billion or $11,900 per person per year.17 IBD includes Crohn's Disease (CD) and Ulcerative Colitis (UC). While these diseases are collectively referred as IBD, there are distinct differences - most notably the area of the intestinal tract affected and the extent of the inflammation. UC typically affects the colon; the disease usually starts at the anus and may progress upward, and may even involve the entire colon. While in CD, the inflammation tends to occur in patches and may involve any area throughout the entire intestinal tract; however, it most often affects the terminal ileum of the small intestine. Inflammation due to UC involves only the inner intestinal mucosa, while the inflammation in CD disease can extend through the entire thickness of the bowel wall.

The management of CD is challenging due to extra-intestinal manifestations and overlapping symptomology with other inflammatory disorders. Treatment typically targets symptom relief, but and patients' ability to tolerate therapy also plays a key role. UC is characterized by lifelong relapsing and remitting colorectal inflammation. The cause of UC is unknown, but is thought to result from an aberrant immune response to environmental factors in genetically predisposed individuals. Metagenomic studies have shown that both patients with UC and recurrent Clostridiodes difficile infection (rCDI) lack diversity and richness of their colonic microbiota and remain in a state of chronic dysbiosis. While current drug treatments and surgery to remove the colon and rectum can reduce symptoms, they are costly, associated with adverse effects, and do not promote the restoration of healthy gut bacteria. Recent studies have shown that fecal microbiota transplant (FMT) is effective in treating IBD. Recent trials in both CD and UC patients have shown FMT to be an effective therapy to induce and maintain clinical remission.

Microscopic colitis (MC) is a chronic inflammatory disease of the colon as manifested by chronic, watery, non-bloody diarrhea. MC usually occurs in middle-aged individuals with a female preponderance. Currently, there are limited treatment options for MC; budesonide may be effective for short-term treatment of MC and can improve quality of life. However, up to 80% will experience symptomatic relapse following cessation of budesonide. Routine maintenance treatment with budesonide is controversial as long-term treatment may increase the risk of steroid-related side effects.

IBS is characterized by chronic, relapsing abdominal discomfort and altered bowel movements - constipation, diarrhea or mixed (diarrhea and constipation). IBS affects approximately 15-20% of Canadians and its economic and social burden is estimated to be over $6.5 billion per year in healthcare costs, work productivity losses, and reduced quality of life (QoL). The etiology and pathophysiology of IBS are not yet established, but appear to be a complex interplay between the host and environment factors. Currently, there are no evidence-based therapies available to cure IBS. Studies have shown that fecal microbiota transplantation (FMT) may be an effective treatment IBS. Given the lack of safe and effective treatment for IBD and IBS which are thought to be due to gastronintestinal dysbiosis, this study was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Able to provide informed consent.
* Willing and able to comply with all the required study procedures.
* Rectally colonized with antimicrobial resistant organisms: Extended-spectrum of beta-lactamase, Carbapenem resistant, vancomycin resistant enterococci

Exclusion Criteria:

* Planned or actively taking another investigational product
* Patients with neutropenia with absolute neutrophil count <0.5 x 109/L
* Evidence of toxic megacolon or gastrointestinal perforation on abdominal x-ray
* Peripheral white blood cell count > 30.0 x 109/L AND temperature > 38.0 ºC
* Active gastroenteritis due to Salmonella, Shigella, shiga toxin-producing E. coli, Yersinia or Campylobacter.
* Unable to tolerate FMT or enema for any reason.
* Requiring systemic antibiotic therapy at the time of FMT.
* Actively taking Saccharomyces boulardii or other probiotic; yogurt is allowed
* Severe underlying disease such that the patient is not expected to survive for at least 30 days.
* History of severe allergy to any food

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, Principal Investigator — Vancouver Island Health Authority
Locations (1):
- Vancouver Island Health Authority, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with IBD or IBS were recruited to receive FMT via rectal administration in the outpatient medical clinic.
Period: Overall Study
Arm/Group | Open Label
Started | 33
Completed | 21
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 33 participants were enrolled for this study. 11 had ulcerative colitis 16 had irritable bowel syndrome 3 had Crohn's disease 3 had microscopic colitis
  years
    Ulcerative colitis: number analyzed (Participants) | 11
    Ulcerative colitis | 36.36 (12.06)
    Irritable bowel syndrome: number analyzed (Participants) | 16
    Irritable bowel syndrome | 52.94 (15.20)
    Crohn's disease: number analyzed (Participants) | 3
    Crohn's disease | 46.33 (9.45)
    Microscopic colitis: number analyzed (Participants) | 3
    Microscopic colitis | 54.67 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 33 participants were enrolled for this study. 11 had ulcerative colitis 16 had irritable bowel syndrome 3 had Crohn's disease 3 had microscopic colitis
  Participants
    Ulcerative colitis: number analyzed (Participants) | 11
    Ulcerative colitis: Female | 7
    Ulcerative colitis: Male | 4
    Irritable bowel syndrome: number analyzed (Participants) | 16
    Irritable bowel syndrome: Female | 9
    Irritable bowel syndrome: Male | 7
    Crohn's disease: number analyzed (Participants) | 3
    Crohn's disease: Female | 1
    Crohn's disease: Male | 2
    Microscopic colitis: number analyzed (Participants) | 3
    Microscopic colitis: Female | 3
    Microscopic colitis: Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 33 participants were enrolled for this study. 11 had ulcerative colitis 16 had irritable bowel syndrome 3 had Crohn's disease 3 had microscopic colitis
  Participants
    Ulcerative colitis: number analyzed (Participants) | 11
    Ulcerative colitis: American Indian or Alaska Native | 0
    Ulcerative colitis: Asian | 1
    Ulcerative colitis: Native Hawaiian or Other Pacific Islander | 0
    Ulcerative colitis: Black or African American | 0
    Ulcerative colitis: White | 10
    Ulcerative colitis: More than one race | 0
    Ulcerative colitis: Unknown or Not Reported | 0
    Irritable bowel syndrome: number analyzed (Participants) | 16
    Irritable bowel syndrome: American Indian or Alaska Native | 0
    Irritable bowel syndrome: Asian | 0
    Irritable bowel syndrome: Native Hawaiian or Other Pacific Islander | 0
    Irritable bowel syndrome: Black or African American | 0
    Irritable bowel syndrome: White | 16
    Irritable bowel syndrome: More than one race | 0
    Irritable bowel syndrome: Unknown or Not Reported | 0
    Crohn's disease: number analyzed (Participants) | 3
    Crohn's disease: American Indian or Alaska Native | 0
    Crohn's disease: Asian | 1
    Crohn's disease: Native Hawaiian or Other Pacific Islander | 0
    Crohn's disease: Black or African American | 0
    Crohn's disease: White | 2
    Crohn's disease: More than one race | 0
    Crohn's disease: Unknown or Not Reported | 0
    Microscopic colitis: number analyzed (Participants) | 3
    Microscopic colitis: American Indian or Alaska Native | 0
    Microscopic colitis: Asian | 0
    Microscopic colitis: Native Hawaiian or Other Pacific Islander | 0
    Microscopic colitis: Black or African American | 0
    Microscopic colitis: White | 3
    Microscopic colitis: More than one race | 0
    Microscopic colitis: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 33

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of FMT in Active Ulcerative Colitis
Description: Evaluate the Ulcerative Colitis Disease Activity Index from baseline 4 weeks, 12 weeks and 1 year following FMT using partial-MAYO score. Partial-MAYO is a validated scoring system to determine the activity of UC. it uses three non-invasive components (stool frequency, rectal bleeding and physician's global assessment. Each of the 3 clinical parameters is assigned a score from 0 to 3 according to the clinical evaluation with a total possible score of 9. Higher the score, more severe the disease; score of 0 - 1 is considered in remission; 2 - 4 mild; 5 - 7 moderate; > 7 severe colitis.
Time Frame: 1 year
Population: Baseline partial-MAYO score for UC
Measure: Mean (Standard Deviation); unit: partial-MAYO Score
Groups:
- Baseline Partial-MAYO Score: active UC, partial-MAYO score at baseline prior to receiving FMT
Arm/Group | Baseline Partial-MAYO Score
Number analyzed (Participants) | 11
partial-MAYO Score
  Baseline partial-MAYO score | 4.81 (2.36)
  week 4 post-FMT partial-MAYO score | 2.91 (2.07)
  week 12 post-FMT partial-MAYO score | 2.09 (1.81)
  year 1 post-FMT partial-MAYO score | 2.00 (1.95)

2. Primary Outcome: Efficacy of FMT for Irritable Bowel Syndrome
Description: IBS severity symptom severity score scale (IBS-SSS) from baseline compared to following FMT in participants with irritable bowel syndrome. IBS-SSS is a validated instrument with a scoring system which produces a meaningful value that is both reproducible and sensitive to change. The instrument contains five questions across the following domains: pain; distension; bowel score and quality of life. Each question can generate a score from 0 to 100 using prompted visual analogue scales; the total scores can range from 0 to 500 with a maximum total score of 500. IBS-SSS is mild for scores 75 - 175; moderate 176 - 300 and severe if > 300.
Time Frame: 1 year
Population: IBS patients with ROME IV diagnostic criteria
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Irritable Bowel Syndrome: FMT for irritable bowel syndrome as defined by Rome IV diagnostic criteria
Arm/Group | Irritable Bowel Syndrome
Number analyzed (Participants) | 16
score on a scale
  Baseline IBS severity scoring system (IBS-SSS) | 358.73 (95.09)
  year 1 post-FMT IBS severity scoring system | 136.13 (58.97)

3. Primary Outcome: Efficacy of FMT in Crohn's Disease
Description: The Crohn's Disease Activity Index (CDAI) was measured at baseline and following FMT. CDAI is a validated instrument used in adults with active Crohn's disease. The index consists of eight factors, 2 of which are subjective: stool habits; pain; general well being; features of extra intestinal disease; use of opiates for diarrhea; abdominal mass; hematocrit (hct); and percentage of body weight below standard. Scores range from 0 to ~ 600: > 450 is severe disease; 220 - 450 moderately active disease; 150 - 219 mildly active disease. Clinical remission is defined as a CDAI score <150, clinical response is either a CDAI score <150 or a CDAI reduction of ≥100 from baseline.
Time Frame: 4 weeks
Population: There were no unexpected adverse events during the follow-up period
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Crohn's Disease: Crohn's Disease and adverse events
Arm/Group | Crohn's Disease
Number analyzed (Participants) | 3
score on a scale
  Baseline Mean CDAI score | 201.7 [157 to 257]
  Week 4 CDAI Mean Score | 123 [105 to 142]

4. Primary Outcome: Efficacy of FMT in Microscopic Colitis (MC) Based on Physician's Global Assessment
Description: Physician's global assessment and number of unformed bowel movements per 24 hours were employed at baseline and following FMT to assess response to FMT as these parameters used to determine MC treatment in clinical trials and care.
  For physician's global assessment, lower the score, lesser the disease activity: 0 = no disease activity; 1 = mild activity; 2 = moderate activity; 3 = severe disease activity
Time Frame: Baseline to 4 weeks following FMT
Population: Participants with active microscopic colitis
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 3
score on a scale
  Baseline Mean Physician Global Assessment | 1.67 [1 to 2]
  week 4 Mean Physician Global Assessment | 0.67 [0 to 2]

5. Primary Outcome: Efficacy of FMT in Microscopic Colitis (MC) Based on Number of Unformed Bowel Movements in 24 Hours
Description: Physician's global assessment and number of unformed bowel movements per 24 hours were employed at baseline and following FMT to assess response to FMT as these parameters used to determine MC treatment in clinical trials and care.
Time Frame: Baseline to 4 weeks following FMT
Population: participants with microscopic colitis
Measure: Mean (Full Range); unit: number of unformed bowel movements/24 hr
Groups:
- Efficacy of FMT in Microscopic Colitis Based on Number of Unformed Bowel Movements in 24 Hours: Microscopic colitis disease activity based on physician's global assessment combined with number of unformed bowel movements in 24 hours
Arm/Group | Efficacy of FMT in Microscopic Colitis Based on Number of Unformed Bowel Movements in 24 Hours
Number analyzed (Participants) | 3
number of unformed bowel movements/24 hr
  Baseline mean number of unformed bowel movements in 24 hours | 7 [5 to 10]
  Week 4 mean number of unformed bowel movements in 24 hours | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: Ulcerative colitis and irritable bowel syndrome 1 year. Crohn's disease 4 weeks (2 participants) to 1 year (1 participant). Microscopic colitis 4 weeks (2 participants) to 1 year (1 participant)
Description: Adverse event (AE) data were collected from the time of enrollment to 1 year following the initial FMT for participants with ulcerative colitis and irritable bowel syndrome.
  *AE data were collected from the time of enrollment to 1 year following the initial FMT for 1 participant each in the Crohn's disease and microscopic colitis groups; AE data were collected from the time of enrollment to 4 weeks following initial FMT from 2 participants from these 2 groups
Groups:
- Ulcerative Colitis: Ulcerative colitis and adverse events
  Fecal Microbiota Transplantation: Fecal Microbiota Transplantation Rectal Administration Open Label
- Irritable Bowel Syndrome: Irritable bowel syndrome and adverse events
- Microscopic Colitis: Microscopic Colitis and adverse events
Arm/Group | Ulcerative Colitis | Irritable Bowel Syndrome | Crohn's Disease | Microscopic Colitis
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/16 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/16 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/11 | 0/16 | 0/3 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulcerative Colitis (N=11) | Irritable Bowel Syndrome (N=16) | Crohn's Disease (N=3) | Microscopic Colitis (N=3)
Colitis - colectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
chronic appendicitis - appendectomy (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulcerative Colitis (N=11) | Irritable Bowel Syndrome (N=16) | Crohn's Disease (N=3) | Microscopic Colitis (N=3)
fatigue (General disorders) | 3 (3) | NA | NA | NA

LIMITATIONS AND CAVEATS:
No Individuals with antibiotic resistant organism colonization or pouchitis were enrolled into the study.

In addition, patient-reported Health-Related Quality of Life outcomes via validated questionnaire, RAND were not completed by the participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03834051/Prot_SAP_000.pdf